CLINICAL TRIAL: NCT05599282
Title: A 90-day, Double-blind, Placebo-controlled, Randomized, Parallel-Group Efficacy and Safety Study of an Amino Acid Supplement in Adults
Brief Title: The Efficacy and Safety of an Amino Acid Supplement in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZandA Technologies, llc (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21ZTCPS01
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Insulin-Like Growth Factor I; Healthy
Keywords: Safety and Efficacy; Amino Acid Supplement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Concealment of the allocation of study arms will be employed using opaque sealed envelopes, each labeled with a randomization number. Each envelope will contain information regarding the study arm associated with each randomization number. These envelopes will be readily available for the Qualified Investigator to open in the event that it becomes necessary to know which product a participant is taking for the sake of participant health care.
  Unblinding should not occur except in the case of emergency situations. If a serious adverse event occurs, for which the identity of the investigational product (IP) administered is necessary to manage the participant's condition, the study arm assigned to the participant will be unblinded and the IP identified.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amino Acid Supplement (Experimental): Participants will be instructed to take four (4) capsules of Amino Acid Supplement with a full glass of water daily for up to 90 days, starting on day 1. No substance other than water (i.e., food, drink other than water, and/or medication, supplement, vitamin, and/or mineral) can be consumed two hours before or after taking the Investigational Product (IP). The IP must be consistently consumed immediately before nighttime sleep throughout the study.
  If a dose is missed participants are instructed to record the missed dose in their study journal. Missed doses will not be taken at a later time or date. If any substance other than water is consumed two hours before or after taking the IP, that IP use will be counted as a missed dose. Participants will be advised not to exceed four (4) capsules daily.
  Interventions: Drug: Amino Acid Supplement
- Placebo (Placebo Comparator): Participants will be instructed to take four (4) capsules of Placebo with a full glass of water daily for up to 90 days, starting on day 1. No substance other than water (i.e., food, drink other than water, and/or medication, supplement, vitamin, and/or mineral) can be consumed two hours before or after taking the placebo. The placebo must be consistently consumed immediately before nighttime sleep throughout the study.
  If a dose is missed participants are instructed to record the missed dose in their study journal. Missed doses will not be taken at a later time or date. If any substance other than water is consumed two hours before or after taking the placebo, that placebo use will be counted as a missed dose. Participants will be advised not to exceed four (4) capsules daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amino Acid Supplement — Four capsules of Amino Acid Supplement will be taken once a day for 90 days.
  Arms: Amino Acid Supplement
Other: Placebo — Four capsules of Placebo will be taken once a day for 90 days.
  Arms: Placebo

SUMMARY:
The primary objective of this clinical trial is to determine the efficacy of once daily oral AAS use, as compared to placebo, in increasing serum IGF-1 concentrations within adults aged 35-75 years for up to 90 days. Additionally, the safety and tolerability of the AAS, as compared to placebo, will be measured by the occurrence of and/or changes in treatment-emergent adverse events (AEs).

For the study population, the eligibility criteria limit the presence of confounding variables that could influence study outcomes. Participants will be men and women between 35 and 75 years of age to account for the age range in which humans experience a decline in HGH/IGF-1. Each participant will be deemed eligible to participate by the Qualified Investigator (QI) by means of an extensive review of medical history, laboratory results, and physical examination. Participants will be required to have body mass index (BMI) measurements between 18.5 and 35.0 kg/m2 to ensure that their body weight/composition will not have a confounding effect on their HGH levels (18, 19) and to facilitate generalizability. Participants will be required to maintain current medication and supplements use and sleep throughout the study. They must also abstain from any over-the counter (OTC) medications and/or supplements that may affect the efficacy or safety of the AAS.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 35-75 years of age at baseline
2. Weigh at least 52 kg for males and 45 kg for females
3. BMI between 18.5-35.0 kg/m2, inclusive at screening
4. Serum IGF-1 concentrations within ≤ 2 SDs of age-adjusted reference range as defined by the clinical laboratory
5. Individual is not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
6. Provided voluntary, written, informed consent to participate in the study.
7. Agrees to maintain current lifestyle habits throughout the study, including medications, supplements, and sleep.
8. Agrees to avoid taking new supplements.
9. Willingness to complete study assessments, journals, and all clinic visits
10. Deemed eligible to participate as determined by medical history, laboratory results, and physical exam as assessed by QI

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to investigational product (IP) and/or placebo active or inactive ingredients
3. Has a condition known to directly involve and/or affect IGF-1, including acromegaly, dwarfism, malnutrition, pituitary disorders, and Laron Syndrome
4. Current or history of any significant diseases involving dementia (e.g., Alzheimer's disease, vascular dementia, etc.)
5. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable.
6. Current diagnosis or history of chronic kidney disease (creatinine levels > 1.1 mg/dl for women; > 1.2 mg/dl for men)
7. Current diagnosis or history of a thyroid-related disorder and/or disease
8. Current diagnosis of liver diseases
9. Current diagnosis of primary hypercholesterolemia (LDL-C 160-189 mg/dl [4.1-4.8 mmol/l]; non-HDL-C 190-219 mg/dl [4.9-5.6 mmol/l])
10. Current diagnosis of primary hypertriglyceridemia (triglycerides >150 mg/dl, fasting)
11. Current diagnosis of stage 2 hypertension (> 140/90 mmHg)
12. Current diagnosis of type 1 or type 2 diabetes mellitus (HbA1c > 6.5%)
13. History or presence of gastrointestinal (including prior bariatric bypass surgery), hepatic or renal disease, or any other condition that may interfere with the absorption, distribution, metabolism, or excretion of IPs, based on the opinion of the QI
14. History of cardiovascular disease and/or significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
15. History (within past two years at screening) or presence of diagnosis of alcohol abuse, a substance abuse disorder, known drug dependence, or seeking treatment for alcohol or substance abuse related disorder.
16. Current use of prescribed medications, over-the-counter (OTC) medications, or supplements which may affect the efficacy and/or safety of the IP
17. Individuals who work or plan to work night shifts
18. Individuals who have travelled to other time zones within two weeks prior to baseline or plan to travel to other time zones during the study
19. Alcohol intake average of > 2 standard drinks per day as assessed by the QI
20. Clinically significant abnormal laboratory results at screening as assessed by the QI
21. Participation in other clinical research studies 30 days prior to enrollment will be assessed on a case-by-case basis by the QI
22. Individuals who are unable to give informed consent
23. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
The difference in serum IGF-1 concentrations from baseline up to 30 days of supplementation between Amino Acid Supplement (AAS) compared to placebo. | baseline (day 1) and 31 days
  The difference in serum IGF-1 concentrations (ng/ml) from baseline (day 1) to 30 days (day 31) of supplementation between AAS will be compared to placebo
The difference in serum IGF-1 concentrations from baseline up to 60 days of supplementation between Amino Acid Supplement (AAS) compared to placebo. | baseline (day 1) and 61 days
  The difference in serum IGF-1 concentrations (ng/ml) from baseline (day 1) up to 60 days (day 61) of supplementation between AAS will be compared to placebo
The difference in serum IGF-1 concentrations from baseline up to 90 days of supplementation between Amino Acid Supplement (AAS) compared to placebo. | baseline (day 1) and 91 days
  The difference in serum IGF-1 concentrations (ng/ml) from baseline (day 1) up to 90 days (day 91) of supplementation between AAS will be compared to placebo

SECONDARY OUTCOMES:
Incidence of pre-emergent adverse events following 90 days of supplementation with Amino Acid Supplement (AAS) compared to placebo | 105 days
  Incidence of pre-emergent adverse events following 90 days of supplementation with Amino Acid Supplement (AAS) will be compared to placebo. A follow-up safety call will also be conducted 2 weeks after the 90 day treatment (day 105) with Amino Acid Supplement.
Incidence of post-emergent adverse events following 90 days of supplementation with Amino Acid Supplement (AAS) compared to placebo | 105 days
  Incidence of post-emergent adverse events following 90 days of supplementation with Amino Acid Supplement (AAS) will be compared to placebo. A follow-up safety call will also be conducted 2 weeks after the 90 day treatment (day 105) with Amino Acid Supplement.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada